CLINICAL TRIAL: NCT03151135
Title: Does Energy Turnover After Short-term Nutritional Recovery Predict Subsequent Weight Course in Patients With Anorexia Nervosa?
Brief Title: Energy Turnover in Patients With Anorexia Nervosa
Status: Terminated | Type: Observational
Why Stopped: Funding period expired before all subjects could be recrutied
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Research Foundation (Other); Hannover Medical School (Other); Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Dr. Verena Haas, Dr. oec. troph. Verena Haas, PhD, Charite University, Berlin, Germany
Other Study IDs: DLW_AN
Record Dates: First submitted 2017-04-07; First posted 2017-05-12 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Anorexia Nervosa
Keywords: Energy metabolism
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AN patients: Patients with Anorexia Nervosa (AN). No intervention, observation at end of inpatient treatment

SUMMARY:
Pilot study to assess energy turnover at end of inpatient treatment in 10 patients with Anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Anorexia nervosa
* anabolic metabolism
* high compliance
* end of inpatient treatment

Exclusion Criteria:

* any further disease than eating disorder
* smokers

Ages: 13 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Anorexia nervosa
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Resting Energy expenditure (REE; kcal/d); Total Daily Energy Expenditure (TDEE; kcal/d) | End of inpatient treatment (T0), within 2 weeks before discharge
  REE will be measured in a Respiration chamber and TDEE with isotope dilution

SECONDARY OUTCOMES:
Body weight | T1 = 6 months after first test (T0)
  Body weight 6 months after discharge from inpatient Treatment (T1)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité-Universitätsmedizin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided